CLINICAL TRIAL: NCT01057043
Title: Randomised Controlled Clinical Trial on Pulsatile Cupping in Patients With Osteoarthritis of the Knee.
Brief Title: Cupping in Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Company HeVaTech (Unknown)
Responsible Party: Principal Investigator, Benno Brinkhaus, Prof. MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAI /230/09
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waiting list (No Intervention): In case of acute pain patients may take paracetamol as rescue medication, maximum dosage 2 gram per day.
- Cupping (Experimental): In case of acute pain patients may take paracetamol as rescue medication, maximum dosage 2 gram per day.
  Interventions: Device: Pulsatile cupping

INTERVENTIONS:
Device: Pulsatile cupping — 8 sessions cupping in 4 weeks, administered by a cupping machine. Cupping is administered in each session for 15 minutes with silicon cupping glasses to the knee (osteoarthritis) and the lower back.
  Other Names: Cupping machine: Puls Reguliertes Vakuum PRV 02; HeVaTec ; registered and certified in Germany [MPG] DIMDI Identifizierungscode DE/0000042259)
  Arms: Cupping

SUMMARY:
The purpose of this exploratory randomised trial is to study the effect of pulsatile cupping in osteoarthritis of the knee compared to waiting list control.

DETAILED DESCRIPTION:
Cupping is a traditional therapy in many cultures of the world and is used to treat osteoarthritis of the knee. In this randomised trial we want to study the effect of pulsatile cupping in osteoarthritis of the knee compared to waiting list control. Pulsatile cupping is administered by a special cupping machine (HeVaTec) with silicone cupping glasses to the knee joint. Pulsatile pressure is generated by a pump that generates vacuum.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee according ACR-criteria
* X-ray classification minimum Kellgren-Lawrence criteria grade 2
* Pain Intensity > 40 mm VAS
* Only therapy with NSAIDin the last 4 weeks
* Informed consent

Exclusion Criteria:

* Use of anticoagulants (Phenprocoumon, Heparin)
* Coagulopathy
* Cupping in the last 12 months
* Intraarticular injection of corticosteroids or NSAID into the knee joint in the last 4 months
* Use of systemic corticosteroids in the last 4 weeks
* Physical therapy, leeches or acupuncture in the last 4 months
* Other CAM therapies for the osteoarthritis in the last 4 weeks
* Arthroscopy of the knee joint in the last 12 months
* Paracetamol allergy or intolerance

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis (WOMAC) - Score | 4 weeks

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis (WOMAC) - Scores | 12 weeks
Pain Intensity (Visual Analogue Scale; no pain=0; maximum pain=100 mm) | week 4 and 12
Quality of Life (SF 36) | 4 and 12 weeks
Adverse events and serious adverse events | continously
Global assessment of efficacy by patients | week 4 and 12
Use of rescue medication (paracetamol) | weeks 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Benno Brinkhaus, Professor, MD, Principal Investigator — Charité University Berlin
Locations (1):
- Institiute for Social Medicine, Epidemiology and Health Economy, Charité University Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Teut M, Kaiser S, Ortiz M, Roll S, Binting S, Willich SN, Brinkhaus B. Pulsatile dry cupping in patients with osteoarthritis of the knee - a randomized controlled exploratory trial. BMC Complement Altern Med. 2012 Oct 12;12:184. doi: 10.1186/1472-6882-12-184. PMID 23057611